CLINICAL TRIAL: NCT02130284
Title: In-Clinic Evaluation of the Predictive Low Glucose Management (PLGM) System in Adult and Pediatric Insulin Requiring Patients With Diabetes Using the Enlite 3 Sensor
Brief Title: In Clinic Evaluation of the PLGM Feature
Acronym: PLGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 272 PLGM
Record Dates: First submitted 2014-04-18; First posted 2014-05-05 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Predictive Low Glucose Management (PLGM) (Experimental): To evaluate the safety of the Predictive Low Glucose Management feature in insulin pump algorithm with the Enlite 3 Sensor
  Interventions: Device: Predictive Low Glucose Management Feature in Insulin pump

INTERVENTIONS:
Device: Predictive Low Glucose Management Feature in Insulin pump — All subjects will undergo hypoglycemic induction at Visit 2 with target set to 65 mg/dL using the rate of change basal increase algorithm. Low Limit setting when PLGM ON is 65 mg/dL.
  Other Names: Medtronic MiniMed 640G Insulin Pump, MMT-1512

SUMMARY:
This study is a multi-center, single arm and in-clinic study to evaluate the safety of the PLGM System and its algorithm with the Enlite 3 Sensor.

DETAILED DESCRIPTION:
A total of up to 95 subjects with type 1 diabetes (age 14-75 years old) will be enrolled at up to 8 investigational centers in order to reach a minimum of 60 subjects who will complete the study (N=minimum 40 adult subjects, 22-75 years old) and N=minimum 15 pediatric subjects (14-21 years old). Subjects will be evaluated in an in-clinic setting with induction of hypoglycemia by increasing their basal rate using a standardized titration tool referred to in protocol as rate of change basal increase algorithm (Buckingham, Diabetes Care 5, 2010). Total duration of frequent sample testing (FST) using Yellow Springs Instrument (YSI) may be up to 19 hours.

Subjects will undergo in-clinic testing on Sensor Day 1.

All subjects will undergo hypoglycemic induction at Visit 2 with target set to 65 mg/dL using the rate of change basal increase algorithm. Low Limit setting when PLGM ON is 65 mg/dL.

The In-Clinic part of the study consists of hypoglycemic induction and an observation period.

Hypoglycemic induction ends when one of the following 3 criteria is met, whichever comes first:

1. PLGM is activated
2. YSI glucose is less than or equal to 65 mg/dL, followed by the next YSI sample less than or equal to 65 mg/dL (2 contiguous YSI samples).
3. Neither condition for #1 or #2 has been met in 12 hours

Observation with YSI ends when:

1. If PLGM is activated, observation with YSI frequent sample testing will include the Suspend period (30 minutes minimum to 2 hours maximum) and insulin resumption period (approximately 4 hours from the time insulin delivery resumes). This may include insulin re-suspension during this period. Maximum observation with YSI frequent sample testing should be no longer than 19 hours.
2. YSI glucose less than or equal to 65 mg/dL is followed by the next YSI sample less than or equal to 65 mg/dL (2 contiguous YSI samples). The subject will be rescued and YSI observation will end
3. Twelve hours have passed since the start of hypoglycemic induction without PLGM activation
4. See In-Clinic Stopping rules

Enrollment for this study will proceed in phases.

Phase 1 only allows enrollment of adult subjects (22-75 years). Subjects will wear pump system, as shown below:

* One Study Pump
* One GST-3C Transmitter
* One Enlite 3 Sensor

Progression to Phase 2 may occur after 10 adult subjects have completed Phase 1 and a Data Safety Monitoring Board (DSMB) has approved that it is safe to continue on to Phase 2.

Phase 2 enrollment involves a minimum of 15 pediatric subjects (14-21). Subjects will wear the same pump system as shown for Phase 1.

A total of up to 95 subjects will be enrolled at up to 10 investigational centers in order to reach a minimum of 60 subjects (N=minimum 40 adult subjects and N=minimum 15 pediatric subjects) who will complete the study.

Considering around 15% screen failure rate and approximately 15% drop-out rate, a total of up to 95 subjects will be enrolled in order to have 60 subjects complete the study.

1. The investigational centers will be encouraged to include subjects of different ethnicities including Hispanic, Native American, and African-American
2. Subjects will be grouped into cohorts by Age

The study is anticipated to last no longer than 12 months from investigational center initiation to completion of all data entry and monitoring procedures including final report. Subjects can expect to participate for approximately 2-3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 14-75 years of age at time of screening
2. Subject has a clinical diagnosis of type 1 diabetes, as determined via medical record or source documentation by an individual qualified to make a medical diagnosis

   Inclusion Criteria that are Based on Demands of In-Clinic Study Procedures
3. On pump therapy at the time of screening with insulin sensitivity and insulin carbohydrate ratio
4. Adequate venous access as assessed by investigator or appropriate staff

Exclusion Criteria:

Exclusion Criteria that are Based on Demands of In-Clinic Study Procedures

1. Subject is unable to tolerate tape adhesive in the area of sensor placement
2. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject has a positive urine or serum pregnancy screening test
5. Subject is female, sexually active without use of contraception and plans to become pregnant during the course of the study
6. Subject has had a hypoglycemic induced seizure within the past 6 months prior to screening visit
7. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit
8. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit
9. Subject has a history of a seizure disorder
10. Subject has central nervous system or cardiac disorder resulting in syncope
11. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
12. Subjects with hematocrit (Hct) lower than the normal reference range for age per local lab testing
13. Subjects with a history or findings on screening electrocardiogram (EKG) of any cardiac arrhythmia, including atrial arrhythmias
14. Subjects with a history of adrenal insufficiency
15. Subjects with history of migraines that have occurred at least 2 times in the last 3 months prior to enrollment

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, MD, Study Director — Medtronic Diabetes
Locations (8):
- United States (8):
  - AMCR Institute, Inc., Escondido, California
  - Stanford University Department of Pediatric Endocrinology, Stanford, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center of Childhood Diabetes, Denver, Colorado
  - Yale University Diabetes Research Program, New Haven, Connecticut
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - University of Virgina, Charlottesville, Virginia
  - Rainier Clinical Research, Renton, Washington

REFERENCES:
- [Derived] Buckingham BA, Bailey TS, Christiansen M, Garg S, Weinzimer S, Bode B, Anderson SM, Brazg R, Ly TT, Kaufman FR. Evaluation of a Predictive Low-Glucose Management System In-Clinic. Diabetes Technol Ther. 2017 May;19(5):288-292. doi: 10.1089/dia.2016.0319. Epub 2017 Feb 16. PMID 28221823

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Predictive Low Glucose Management (PLGM)
Started | 80
Completed | 71
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Subject Withdrew Consent | 1
Not completed — Subject's sensor failed at Visit 2, Day | 1
Not completed — Subject was screened as backup for study | 3
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 63
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (16.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events (SAE)
Description: Evaluation of incidence of SAE during in-clinic procedures
Time Frame: From start of in clinic procedures until the end of the study, which may occur up to 48 hours after the start of in-clinic procedures
Measure: Count of Participants; unit: Participants
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
Participants | 0

2. Primary Outcome: Unanticipated Device Effect (UADE)
Description: Evaluation of incidence of UADE during in-clinic procedures
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
Participants | 0

3. Primary Outcome: Severe Hypoglycemia
Description: Evaluation of incidence of severe hypoglycemia during in-clinic procedures
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
Participants | 0

4. Primary Outcome: Diabetic Ketoacidosis
Description: Evaluation of DKA during in-clinic procedures
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
Participants | 0

5. Primary Outcome: Rescue Events During In-clinic Procedues
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
Participants | 7

6. Other Pre Specified Outcome: PLGM Performance - Hypoglycemia Event Rate at Threshold of YSI <= 65 mg/dL.
Description: Hypoglycemic event rate among 71 subjects who underwent the PLGM experiment. Hypoglycemic events are defined based on: occurrence of 2 or more continuous YSI <= 65 mg/dL during in-clinic procedures.
Time Frame: as for outcome 1
Population: Two subjects were excluded from analysis because the site staff did not set the pump up correctly prior to YSI and the PLGM feature was never set to activate.
Measure: Number; unit: percentage of total subjects
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 69
percentage of total subjects | 39.13

7. Other Pre Specified Outcome: Sensor Performance: Accuracy
Description: MARD (Mean Absolute Relative Difference) between sensor glucose value and YSI. MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100).
Time Frame: as for outcome 1
Population: Total of 71 subjects completed the study. However, two subjects who withdrew also had YSI and Sensor glucose values. Therefore, total of 73 subjects contributed to sensor accuracy analysis
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 73
percentage | 12.56 (10.06)

8. Other Pre Specified Outcome: Device Metric/Performance - All Device Deficiencies
Time Frame: as for outcome 1
Measure: Number; unit: device performance issues
Arm/Group | Predictive Low Glucose Management (PLGM)
Number analyzed (Participants) | 80
device performance issues | 13

ADVERSE EVENTS:
Arm/Group | Predictive Low Glucose Management (PLGM)
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 5/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Predictive Low Glucose Management (PLGM) (N=80)
Upper respiratory infection (Infections and infestations) | 1 (1)
Mild back strain (Injury, poisoning and procedural complications) | 1 (1)
emesis (Gastrointestinal disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days